CLINICAL TRIAL: NCT05698680
Title: Pragmatic, Randomized, Multicenter, Double-blind, Controlled, Clinical Trial of Prednisolone Versus Colchicine for Acute Gout in Primary Care
Brief Title: Prednisolone Versus Colchicine for Acute Gout in Primary Care
Acronym: COPAGO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: University of Göttingen (Other); Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202102COPAGO; 01KG2022 (Other Grant/Funding Number: German Federal Ministry of Education and Research); 2024-514738-18-00 (EU CTIS Number); 2021-005556-11 (EudraCT Number)
Record Dates: First submitted 2022-12-27; First posted 2023-01-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Acute Gout
Keywords: Primary care; Prednisolone; Colchicine; Pragmatic
MeSH Terms: interventions — Prednisolone; Tablets; Colchicine

STUDY DESIGN:
Intervention Model Description: This clinical trial is a two-arm multicentre, pragmatic, prospective, randomised, double-blind, controlled clinical trial of prednisolone and colchicine for non-inferiority with a parallel group design (phase IV).
  According to the guidelines of the German Society of General Medicine (DEGAM), the decision to start gout treatment is made clinically. As this is a pragmatic study, eligibility will be determined during a routine clinical examination. The clinical diagnosis is made without new laboratory tests, joint puncture with synovial analysis or imaging.
  314 patients with an acute gout attack are going to be recruited in 60 General Practitioner's practices across 3 university sites (Greifswald, Göttingen, and Würzburg). All study participants receive active treatments, but are randomised into either the prednisolone group (treatment group) or the colchicine group (comparison group). The study lasts 4 weeks for each participant.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There are 2 active and effective treatments (colchicine vs. prednisolone). The allocation to the treatment arms is 1:1, and study participants are randomised to either group. Randomisation is intended to reduce selection and allocation bias.
  As both drugs have different dosing regimens, the investigators provide identical blisters for both drugs including the active substance and corresponding placebos. This way, all study participants receive the same number of tablets and the possibility of drug prediction is more difficult. This is achieved by using tablets that are identical in taste and appearance (double-dummy design). Participants randomised to the colchicine arm will receive colchicine plus prednisolone placebo. Participants randomised to the prednisolone arm will receive prednisolone plus a colchicine placebo. The prednisolone placebos contain a bittering agent due to the bitter taste of prednisolone to ensure a similar taste.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisolone 30mg (Day 0-4) (Experimental): As both drugs have different dosing regimens, the investigators provide identical blisters for both drugs including the active substance and corresponding placebos. This way, all study participants receive the same number of tablets and the possibility of drug prediction is more difficult. This is achieved by using tablets that are identical in taste and appearance (double-dummy design). Participants randomised to the prednisolone arm will receive prednisolone plus a colchicine placebo. The prednisolone placebos contain a bittering agent due to the bitter taste of prednisolone to ensure a similar taste.
  The dosage is according to EULAR guideline and also within the recommended range of the DEGAM guideline. The cumulative total dose taken per participant within the clinical trial is 150 mg for prednisolone.
  Interventions: Drug: Prednisolone 30 mg Tablet
- Colchicine 1.5 mg (Day 0), 1.0 mg (Day 1-4) (Active Comparator): As both drugs have different dosing regimens, the investigators provide identical blisters for both drugs including the active substance and corresponding placebos. This way, all study participants receive the same number of tablets and the possibility of drug prediction is more difficult. This is achieved by using tablets that are identical in taste and appearance (double-dummy design). Participants randomised to the colchicine arm will receive colchicine plus prednisolone placebo.
  The dosage is according to EULAR guideline and also within the recommended range of the DEGAM guideline. The cumulative total dose taken per participant within the clinical trial is 5.5mg for colchicine.
  Interventions: Drug: Colchicine 0.5 mg Oral Tablet

INTERVENTIONS:
Drug: Prednisolone 30 mg Tablet — See treatment arm "Prednisolone"
  Other Names: + Placebo
  Arms: Prednisolone 30mg (Day 0-4)
Drug: Colchicine 0.5 mg Oral Tablet — See treatment arm "Colchicine"
  Other Names: + Placebo
  Arms: Colchicine 1.5 mg (Day 0), 1.0 mg (Day 1-4)

SUMMARY:
Gout is the most common form of rheumatic disease in which monosodium urate crystals are deposited in the joints followed by acute inflammatory reactions. There are various approved drugs that can be prescribed for pain relief during an acute gout attack. However to date, no direct comparison of efficacy of colchicine and prednisolone for the treatment of acute gout attacks has been investigated. Furthermore, majority of previous research studies were not only conducted in tertiary centres but also excluded patients with common comorbidities due to contraindications with naproxen.

This pragmatic, prospective, double-blind, parallel-group, randomized, non-inferiority trial will investigate whether prednisolone (treatment drug) is comparable or only acceptably worse than treatment with colchicine (comparison drug) in patients presenting with acute gout. Patients presenting with acute gout to their general practitioners in 60 practices across 3 university sites (Greifswald, Göttingen, and Würzburg) will be invited to participate. Patients often excluded by previous studies due to contraindications with naproxen will also be able to participate. The investigators will compare the absolute levels of the most severe pain on day 3 (in the last 24 hours) measured with an 11-item numerical rating scale as the primary endpoint. Day 0 is the day patients take their study medication for the first time. They are then asked to fill out a study diary at the same time each day to quantify their pain. Pain scores will then be used as comparison between the two medications.

DETAILED DESCRIPTION:
SCIENTIFIC BACKGROUND:

Gout is one of the most common rheumatic diseases, affecting 3-6% of men and 1-2% of women in western countries. Due to the severe pain and impaired quality of life, the individual burden of disease during an acute gout attack is very high. Currently, there are several approved medications available for the treatment of acute gout attacks. The EULAR (European League Against Rheumatism) guideline recommends colchicine as the drug of first choice for acute gout attacks. But according to it, non-steroidal anti-inflammatory drugs (NSAIDs) and systemic corticosteroids can also be used. In contrast, DEGAM (German Society for General Medicine and Family Medicine) recommends using prednisolone.

Most commonly, gout attacks are treated in general practices. However, studies on the treatment of acute gout attacks have so far been conducted mainly in specialised centres, and thus in a selective patient group. The gold standard for the diagnosis of gout in rheumatology centres is the detection of monosodium urate crystals in aspirated joint fluid. In primary care, however, the diagnosis of gout is made on the basis of clinical symptoms alone. Because of the risk of injury and infection, joint puncture is not usually performed on patients in a general practice setting.

Prednisolone and low-dose colchicine were selected for the study due to a high prevalence of patients with contraindications to NSAIDs, including, cardiovascular disease, oral anticoagulation, chronic kidney disease or a history of gastrointestinal disease. Approximately 20-30% of patients with gout are poorly suited for NSAID administration and in previous studies, those patients were excluded.

RESEARCH QUESTION:

This non-inferiority trial is going to investigate whether prednisolone (treatment drug) is comparable or only acceptably worse than treatment with colchicine (comparator drug). Both treatments will be compared on the basis of the absolute pain scores achieved on day 3 of follow-up.

Unlike most studies conducted in tertiary care centres, this study is going to be set in primary care. The dosage of the study's medications will be according to the recommendations of the EULAR and DEGAM guidelines. Both drugs are in tablet form. Since a preference of the treating physicians regarding the use of prednisolone or colchicine is suspected, the study will be conducted in a double-blinded manner. Due to the different intake regimen, placebos will be used in addition to the effective medications (double-dummy method).

DUAL ENERGY COMPUTED TOMOGRAPHY:

The dual energy computed tomography (DECT) is able to detect monosodium urate crystals. The amount of monosodium urate crystals in the joint (volume) is an indicator of disease burden and can also be used to make treatment decisions regarding uric acid-lowering therapy (ULT) to avoid the occurrence of potential future gout attacks. Although imaging techniques, such as DECT, show promise in classifying symptomatic gout, studies to date are small and mainly involve people with long-standing, established disease from a hospital setting. In those with the first acute gout attack, diagnostic sensitivity ranges from 35.7 % to 61.5 %.

Due to the unclear diagnostic sensitivity in first attacks, the DECT examination will not be mandatory in the present study. It will be offered to all participants as optional. About 10% of the participants are expected to have a gout attack in the hand. Since the joints of the feet are the main site of manifestation of acute gout attacks, crystal deposits in the feet are also expected in these study participants. In order to ensure comparability of the volume measurement, the dual energy CT examination is therefore limited to the feet.

The aim of the dual energy CT examination is to describe the frequency and volume of monosodium urate crystals in patients with gout in primary care. In a sensitivity analysis, the primary endpoint in patients with positive DECT findings will be analysed. Furthermore, the association between the duration of gout diagnosis and crystal volume as a marker for disease burden will be investigated. The investigation of the frequency and volume of monosodium urate crystals provides the basis for the design of further studies on the usefulness of DECT for the indication and monitoring of uric acid-lowering therapies in primary care.

STUDY PROCEDURE:

During the study, the participants will attend their General Practitioner's practice twice (baseline and one-off on day 6-8), as well as, an optional visit for a DECT at the university medical centre in the local region (Greifswald or Göttingen; day 7-13) and a one-off telephone interview on day 27-34. The study period for the individual participant will be 4 weeks.

On day 0 (day of first presentation at the general practice), patients with an acute gout attack in the hand or foot present to their general practitioner. If the diagnosis of gout is confirmed and patients are eligible for participation in the study, they will be consented and randomly assigned to one of two treatment groups. While patient group 1 is treated with prednisolone for 5 days, patient group 2 receives colchicine for 5 days. So that neither the patient nor the general practitioner knows the allocation, both treatment groups also receive a placebo (dummy medication). A laboratory test will also be performed to determine serum uric acid levels, as well as, inflammatory markers and renal function. The aim of blood collection and determination of laboratory parameters is to descriptively describe the patient population and to perform subgroup analyses with regard to the primary endpoint.

During days 1 to 6, patients are requested to complete a patient diary. The primary and secondary endpoints (pain, joint swelling, joint tenderness) and, if further analgesia is needed, the use of additional pain medication will be recorded in the diary. Participants who have a blood pressure monitor will be asked to measure and record their blood pressure daily. On day 6, the patients are also asked to assess potential functional limitations caused by the gout attack and to give a global assessment of the treatment success.

After one week, patients return for their follow-up visit (visit 2) to their general practitioners. They are examined again and are asked to return their study diary and any remaining medication packets.

After 4 weeks, the patients will be contacted by telephone by our study nurses and asked about the clinical course of their gout attack (recurrence of an acute gout attack, further treatment, duration of incapacity to work, adverse events). The telephone call lasts about 15 minutes.

In addition, study participants will receive the optional offer to have a one-time dual-energy CT examination of their feet on days 7-13 to check for the presence of uric acid crystals. Imaging of both feet using a Siemens Dual Source SOMATOM Definition Flash or SOMATOM Force will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age
* Clinical diagnosis of acute attack of gout (symptoms: pain, swelling, tenderness, redness or local hyperthermia).
* Acute pain in hand or foot (podagra, chiragra)
* The onset of pain was no more than 2 days ago (e.g., presentation on Monday afternoon, onset of pain on Saturday morning)
* Willingness to participate in the study and ability to give written informed consent.

Exclusion Criteria:

* Known intolerance or contraindication to either medication
* Known intolerance to the placebo (e.g. lactose intolerance).
* Existing (or less than 2 weeks ago) oral treatment with corticosteroids or colchicine.
* Known chronic kidney disease (CKD stage 4 or greater) or an available value of estimated glomerular filtration rate (eGFR) < 30ml/min/1.73 m².
* Known haematopoietic disorder or available values of platelets < 30,000 µl or leucocytes < 4000 µl, or Hb <5 mmol/l/ or 8 g/dl
* Uncontrolled high blood pressure (systolic blood pressure permanently above 160 mmHg).
* Known liver cirrhosis or severe liver disease or available liver enzymes results (ie. Serum Glutamate Oxalate Transaminase (SGOT) and Serum Glutamic Pyruvic Transaminase(SGPT)) being elevated by more than twice the respective reference range
* Known current gastric or duodenal ulcer (diagnosed in the last 4 weeks)
* Current chemotherapy or chemotherapy completed less than 3 months ago
* Known HIV infection
* Solid organ transplant with immune suppression
* Desire to have children within the next 6 months in both men and women
* Existing pregnancy or breastfeeding
* Participation in other studies according to the German Medicines Act in the last 3 months
* Participation in the COPAGO study with past gout attack

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Most severe pain in the last 24 hours | Day 3
  To investigate whether the efficacy of prednisolone in General Practitioner's care is equally good or only marginally weaker than treatment with low-dose colchicine, the most severe pain in the last 24 hours on day 3 after baseline on an 11-point numerical rating scale is used and compared across groups. The study participants take their study medication for the first time on day 0 and are then asked to fill out their diary daily at the same time to quantify their pain. 0 stands for no pain and 10 for the strongest pain imaginable.

SECONDARY OUTCOMES:
Average response to treatment | Day 1, 2, 3, 4, 5, 6
  For this purpose, the most severe pain described on an 11-point numerical rating scale across treatment days (from day 1 - 6 of follow-up) is used and compared across groups. The study participants take their study medication for the first time on day 0 and are then asked to fill out their diary daily at the same time to quantify their pain. 0 stands for no pain and 10 for the strongest pain imaginable.
Swelling and tenderness of the joint | Day 3
  Reduction in joint swelling and tenderness measured using 4-point Likert scale on day 3 after baseline per treatment arm, e.g.:
  * Swelling quantified as no joint swelling, palpable, visible, and bulging beyond the joint margins.
  * Sensitivity to touch of the joint is quantified as no pain, pain, pain and winces, and pain, winces and withdraws,
  and subsequent comparison.
Physical function | Day 1 and 6
  Physical function on day 6 compared to baseline will be assessed with the following questions:
  * How much are you now restricted in your normal daily activities by the gout attack?
  * How much trouble do you have putting on a shoe today?
  * How much pain do you have when you walk today?
  * How much trouble do you have grasping and holding something with your affected hand (for example, when unscrewing a bottle)?
  All questions will be described on an 11-point numerical rating scale, 0 indicating "not at all/no problem" and 10 indicating "worst pain ever".
Patients' global assessment of treatment success | Day 6
  This is going to be measured measured with 5-point Likert scale (excellent, very good, good, fair, poor) on day 6 after baseline and treatment arms will be compared.
Most severe pain in the last 24 hours depending on disease duration | Day 1 and 6
  For this outcome the same model specification as for the primary outcome is applied and the adjustment for age will be substituted with adjustment for disease duration.
Frequency of use of additional pain medication by treatment group | Day 1 - 6
  The frequency of use of additional pain medication per treatment group will be compared.
Frequency of use of non-pharmacological pain therapies | Day 1 - 6
  The frequency of use of non-pharmacological pain therapies per treatment group will be compared.

OTHER OUTCOMES:
Dual Energy Computed Tomography Investigation: Presence of monosodium urate crystals | one assessment during days 7 - 13
  The frequency and volume of monosodium urate crystals (milliliter) in feet joints in patients with gout in primary care will be investigated.
Dual Energy Computed Tomography Investigation: Patient characteristics | one assessment during days 7 - 13
  The investigators will investigate the association between the volume of monosodium urate crystals (milliliter) in feet joints and patient characteristics (e.g. age, sex, previous gout attacks).
Dual Energy Computed Tomography Investigation: Use of uricostats and uricosurics | one assessment during days 7 - 13
  The investigators will investigate the association between frequency and volume of monosodium urate crystals (milliliter) in feet joints in patients with gout in primary care and (previous) use of uricostats and uricosurics.
Dual Energy Computed Tomography Investigation: Pain intensity | one assessment during days 7 - 13
  The investigators will investigate the association between the volume of monosodium urate crystals (milliliter) in feet joints in patients with gout in primary care and pain intensity at baseline (on an 11-point numerical rating scale).

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Stracke, Principal Investigator — University Medicine Greifswald
Locations (65):
- Germany (65):
  - Arztpraxis Burgtorstr. 2, Ittlingen, Baden-Wurttemberg
  - Hausarztpraxis Neckarsteinacher Str. 22, Neckargemünd, Baden-Wurttemberg
  - Hausarztpraxis Kleinfeldlein 3, Bad Bocklet, Bavaria
  - Hausarztpraxis Kapellenstraße 3, Bad Kissingen, Bavaria
  - Hausarztpraxis Ludwigstraße 18, Bad Kissingen, Bavaria
  - Hausarztpraxis Goethestraße 15 G, Bad Neustadt an der Saale, Bavaria
  - Hausarztpraxis Ahornstraße 1, Bischofsheim, Bavaria
  - Hausarztpraxis Mechenharder Straße 174, Erlenbach am Main, Bavaria
  - Hausarztpraxis Hauptstraße 12, Gössenheim, Bavaria
  - Hausarztpraxis Bahnhofstraße 24, Hammelburg, Bavaria
  - Hausarztpraxis Torgraben 3, Haßfurt, Bavaria
  - Hausarztpraxis Kaiserstraße 43, Kitzingen, Bavaria
  - Hausarztpraxis Rathausstraße 31, Leinach, Bavaria
  - Hausarztpraxis Herrngasse 11 A, Rimpar, Bavaria
  - Hausarztpraxis Spitalstr. 9, Schweinfurt, Bavaria
  - Hausarztpraxis Sulzdorfer Straße 6a, Stadtlauringen, Bavaria
  - Hausarztpraxis Dorfgraben 2a, Würzburg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Hausarztpraxis Moltkestraße 5, Würzburg, Bavaria
  - Hausarztpraxis Point 3, Zellingen, Bavaria
  - Hausarztpraxis Wissmannstraße 14, Bad Lauterberg im Harz, Lower Saxony
  - Hausarztpraxis Hoher Weg 17, Bilshausen, Lower Saxony
  - Hausarztpraxis Bohlendamm 2, Gleichen, Lower Saxony
  - Hausarztpraxis Liererstr. 28, Goslar, Lower Saxony
  - Universitätsmedizin Göttingen, Göttingen, Lower Saxony
  - Hausarztpraxis Ewaldstr. 40a, Göttingen, Lower Saxony
  - Hausarztpraxis Hennebergstr. 14a, Göttingen, Lower Saxony
  - Hausarztpraxis Backhausstraße 21, Göttingen, Lower Saxony
  - Hausarztpraxis Godehardtstraße 26, Göttingen, Lower Saxony
  - Hausarztpraxis Professor-Eberlein-Str. 6, Hannoversch Münden, Lower Saxony
  - Hausarztpraxis Steinstraße 19, Hannoversch Münden, Lower Saxony
  - Hausarztpraxis Vor dem Tore 2, Hardegsen, Lower Saxony
  - Hausarztpraxis Eckert Osteroder Str. 9, Herzberg am Harz, Lower Saxony
  - Hausarztpraxis Poppe Osteroder Str. 9, Herzberg am Harz, Lower Saxony
  - Hausarztpraxis Hauptstraße 34, Krebeck, Lower Saxony
  - Hausarztpraxis Neue Straße 22, Moringen, Lower Saxony
  - Hausarztpraxis Bahnhofstraße 6, Scheden, Lower Saxony
  - Hausarztpraxis Kampstr. 32, Seesen, Lower Saxony
  - Hausarztpraxis Bluthsluster Straße 2, Anklam, Mecklenburg-Vorpommern
  - Hausarztpraxis Am Westhafen 1, Barth, Mecklenburg-Vorpommern
  - Hausarztpraxis Schlossstraße 43, Dargun, Mecklenburg-Vorpommern
  - Krankenhaus Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Hausarztpraxis Am Mühlentor 5, Greifswald, Mecklenburg-Vorpommern
  - Hausarztpraxis Anklamer Straße 66, Greifswald, Mecklenburg-Vorpommern
  - Hausarztpraxis Lange Straße 53, Greifswald, Mecklenburg-Vorpommern
  - Hausarztpraxis Markt 1, Greifswald, Mecklenburg-Vorpommern
  - Hausarztpraxis Ernst-Thälmann-Ring 66, Greifswald, Mecklenburg-Vorpommern
  - Hausarztpraxis Schulstraße 1a, Groß Kiesow, Mecklenburg-Vorpommern
  - Hausarztpraxis Pommersche Straße 18, Gützkow, Mecklenburg-Vorpommern
  - Hausarztpraxis Prohner Straße 43, Klausdorf, Mecklenburg-Vorpommern
  - Hausarztpraxis August-Levin-Straße 22c, Loitz, Mecklenburg-Vorpommern
  - Hausarztpraxis Bahnhofstraße 16, Lübstorf, Mecklenburg-Vorpommern
  - Hausarztpraxis Oberreihe 41, Lühmannsdorf, Mecklenburg-Vorpommern
  - Hausarztpraxis Juri-Gagarin-Ring 24, Neubrandenburg, Mecklenburg-Vorpommern
  - Hausarztpraxis Störstraße 2, Plate, Mecklenburg-Vorpommern
  - Hausarztpraxis Werdohler Straße 3, Stavenhagen, Mecklenburg-Vorpommern
  - Hausarztpraxis Marienstraße 2-4, Stralsund, Mecklenburg-Vorpommern
  - Hausarztpraxis Dorfstraße 57, Trent, Mecklenburg-Vorpommern
  - Hausarztpraxis Birkenweg 5, Trinwillershagen, Mecklenburg-Vorpommern
  - Hausarztpraxis Otto-Lilienthal-Straße 3, Trollenhagen, Mecklenburg-Vorpommern
  - Hausarztpraxis Ueckerstraße 48, Ueckermünde, Mecklenburg-Vorpommern
  - Hausarztpraxis Lange Straße 55, Waren, Mecklenburg-Vorpommern
  - Hausarztpraxis Wilhelmstraße 3, Wolgast, Mecklenburg-Vorpommern
  - Hausarztpraxis Lambertweg 6, Höxter, North Rhine-Westphalia
  - Hausarztpraxis Straße der Einheit 56, Uder, Thuringia

IPD SHARING:
Plan to Share IPD: Yes
Original data of the analyses will be made available for re-use.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Richter A, Truthmann J, Hummers E, Pereira JFM, Gagyor I, Schuster F, Witte A, Bohm S, Greser A, Kamin P, Stracke S, Dorr M, Bulow R, Engeli S, Chenot JF, Ittermann T. Prednisolone Versus Colchicine for Acute Gout in Primary Care: statistical analysis plan for the pragmatic, multicenter, randomized, and double-blinded COPAGO non-inferiority trial. Trials. 2024 Apr 3;25(1):229. doi: 10.1186/s13063-024-08066-0. PMID 38570873
- [Background] Truthmann J, Freyer Martins Pereira J, Richter A, Schuster F, Witte A, Bohm S, Greser A, Kamin P, Stracke S, Dorr M, Bulow R, Engeli S, Gagyor I, Hummers E, Chenot JF. Prednisolone Versus Colchicine for Acute Gout in Primary Care (COPAGO): protocol for a two-arm multicentre, pragmatic, prospective, randomized, double-blind, controlled clinical trial of prednisolone and colchicine for non-inferiority with a parallel group design. Trials. 2023 Oct 5;24(1):643. doi: 10.1186/s13063-023-07666-6. PMID 37798801
- [Background] Dalbeth N, Merriman TR, Stamp LK. Gout. Lancet. 2016 Oct 22;388(10055):2039-2052. doi: 10.1016/S0140-6736(16)00346-9. Epub 2016 Apr 21. PMID 27112094
- [Background] Campion EW, Glynn RJ, DeLabry LO. Asymptomatic hyperuricemia. Risks and consequences in the Normative Aging Study. Am J Med. 1987 Mar;82(3):421-6. doi: 10.1016/0002-9343(87)90441-4. PMID 3826098
- [Background] Fisher MC, Rai SK, Lu N, Zhang Y, Choi HK. The unclosing premature mortality gap in gout: a general population-based study. Ann Rheum Dis. 2017 Jul;76(7):1289-1294. doi: 10.1136/annrheumdis-2016-210588. Epub 2017 Jan 25. PMID 28122760
- [Background] ten Klooster PM, Vonkeman HE, Voshaar MA, Bode C, van de Laar MA. Experiences of gout-related disability from the patients' perspective: a mixed methods study. Clin Rheumatol. 2014 Aug;33(8):1145-54. doi: 10.1007/s10067-013-2400-6. PMID 24077900
- [Background] Richette P, Doherty M, Pascual E, Barskova V, Becce F, Castaneda-Sanabria J, Coyfish M, Guillo S, Jansen TL, Janssens H, Liote F, Mallen C, Nuki G, Perez-Ruiz F, Pimentao J, Punzi L, Pywell T, So A, Tausche AK, Uhlig T, Zavada J, Zhang W, Tubach F, Bardin T. 2016 updated EULAR evidence-based recommendations for the management of gout. Ann Rheum Dis. 2017 Jan;76(1):29-42. doi: 10.1136/annrheumdis-2016-209707. Epub 2016 Jul 25. PMID 27457514
- [Background] van Echteld I, Wechalekar MD, Schlesinger N, Buchbinder R, Aletaha D. Colchicine for acute gout. Cochrane Database Syst Rev. 2014 Aug 15;(8):CD006190. doi: 10.1002/14651858.CD006190.pub2. PMID 25123076
- [Background] Finkelstein Y, Aks SE, Hutson JR, Juurlink DN, Nguyen P, Dubnov-Raz G, Pollak U, Koren G, Bentur Y. Colchicine poisoning: the dark side of an ancient drug. Clin Toxicol (Phila). 2010 Jun;48(5):407-14. doi: 10.3109/15563650.2010.495348. PMID 20586571
- [Background] Terkeltaub RA, Furst DE, Bennett K, Kook KA, Crockett RS, Davis MW. High versus low dosing of oral colchicine for early acute gout flare: Twenty-four-hour outcome of the first multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-comparison colchicine study. Arthritis Rheum. 2010 Apr;62(4):1060-8. doi: 10.1002/art.27327. PMID 20131255
- [Background] Engel B, Prautzsch H. [Acute gout in primary care]. 2013. Available from: https://www.awmf.org/uploads/tx_szleitlinien/053_032bl_S1_akute_Gicht_2014-05.pdf
- [Background] van Durme CM, Wechalekar MD, Buchbinder R, Schlesinger N, van der Heijde D, Landewe RB. Non-steroidal anti-inflammatory drugs for acute gout. Cochrane Database Syst Rev. 2014 Sep 16;(9):CD010120. doi: 10.1002/14651858.CD010120.pub2. PMID 25225849
- [Background] Janssens HJ, Janssen M, van de Lisdonk EH, van Riel PL, van Weel C. Use of oral prednisolone or naproxen for the treatment of gout arthritis: a double-blind, randomised equivalence trial. Lancet. 2008 May 31;371(9627):1854-60. doi: 10.1016/S0140-6736(08)60799-0. PMID 18514729
- [Background] McKenzie BJ, Wechalekar MD, Johnston RV, Schlesinger N, Buchbinder R. Colchicine for acute gout. Cochrane Database Syst Rev. 2021 Aug 26;8(8):CD006190. doi: 10.1002/14651858.CD006190.pub3. PMID 34438469
- [Background] Janssens HJEM, Fransen J, Janssen M, Neogi T, Schumacher HR, Jansen TL, Dalbeth N, Taylor WJ. Performance of the 2015 ACR-EULAR classification criteria for gout in a primary care population presenting with monoarthritis. Rheumatology (Oxford). 2017 Aug 1;56(8):1335-1341. doi: 10.1093/rheumatology/kex164. PMID 28431109
- [Background] Dalbeth N, Schumacher HR, Fransen J, Neogi T, Jansen TL, Brown M, Louthrenoo W, Vazquez-Mellado J, Eliseev M, McCarthy G, Stamp LK, Perez-Ruiz F, Sivera F, Ea HK, Gerritsen M, Scire CA, Cavagna L, Lin C, Chou YY, Tausche AK, da Rocha Castelar-Pinheiro G, Janssen M, Chen JH, Cimmino MA, Uhlig T, Taylor WJ. Survey Definitions of Gout for Epidemiologic Studies: Comparison With Crystal Identification as the Gold Standard. Arthritis Care Res (Hoboken). 2016 Dec;68(12):1894-1898. doi: 10.1002/acr.22896. Epub 2016 Oct 28. PMID 27014846
- [Background] Roddy E, Clarkson K, Blagojevic-Bucknall M, Mehta R, Oppong R, Avery A, Hay EM, Heneghan C, Hartshorne L, Hooper J, Hughes G, Jowett S, Lewis M, Little P, McCartney K, Mahtani KR, Nunan D, Santer M, Williams S, Mallen CD. Open-label randomised pragmatic trial (CONTACT) comparing naproxen and low-dose colchicine for the treatment of gout flares in primary care. Ann Rheum Dis. 2020 Feb;79(2):276-284. doi: 10.1136/annrheumdis-2019-216154. Epub 2019 Oct 30. PMID 31666237
- [Background] Richette P, Flipo RN, Patrikos DK. Characteristics and management of gout patients in Europe: data from a large cohort of patients. Eur Rev Med Pharmacol Sci. 2015 Feb;19(4):630-9. PMID 25753881
- [Background] Nyberg F, Horne L, Morlock R, Nuevo J, Storgard C, Aiyer L, Hines DM, Ansolabehere X, Chevalier P. Comorbidity Burden in Trial-Aligned Patients with Established Gout in Germany, UK, US, and France: a Retrospective Analysis. Adv Ther. 2016 Jul;33(7):1180-98. doi: 10.1007/s12325-016-0346-1. Epub 2016 May 26. PMID 27230988
- [Background] Johnson TR. Dual-energy CT: general principles. AJR Am J Roentgenol. 2012 Nov;199(5 Suppl):S3-8. doi: 10.2214/AJR.12.9116. PMID 23097165
- [Background] Dalbeth N, Doyle AJ. Imaging tools to measure treatment response in gout. Rheumatology (Oxford). 2018 Jan 1;57(suppl_1):i27-i34. doi: 10.1093/rheumatology/kex445. PMID 29272513
- [Background] Pascart T, Grandjean A, Capon B, Legrand J, Namane N, Ducoulombier V, Motte M, Vandecandelaere M, Luraschi H, Godart C, Houvenagel E, Norberciak L, Budzik JF. Monosodium urate burden assessed with dual-energy computed tomography predicts the risk of flares in gout: a 12-month observational study : MSU burden and risk of gout flare. Arthritis Res Ther. 2018 Sep 17;20(1):210. doi: 10.1186/s13075-018-1714-9. PMID 30223875
- [Background] Uhlig T, Eskild T, Karoliussen LF, Sexton J, Kvien TK, Haavardsholm EA, Dalbeth N, Hammer HB. Two-year reduction of dual-energy CT urate depositions during a treat-to-target strategy in gout in the NOR-Gout longitudinal study. Rheumatology (Oxford). 2022 Apr 18;61(SI):SI81-SI85. doi: 10.1093/rheumatology/keab533. PMID 34247224
- [Background] Ogdie A, Taylor WJ, Weatherall M, Fransen J, Jansen TL, Neogi T, Schumacher HR, Dalbeth N. Imaging modalities for the classification of gout: systematic literature review and meta-analysis. Ann Rheum Dis. 2015 Oct;74(10):1868-74. doi: 10.1136/annrheumdis-2014-205431. Epub 2014 Jun 10. PMID 24915980
- [Background] Choi HK, Burns LC, Shojania K, Koenig N, Reid G, Abufayyah M, Law G, Kydd AS, Ouellette H, Nicolaou S. Dual energy CT in gout: a prospective validation study. Ann Rheum Dis. 2012 Sep;71(9):1466-71. doi: 10.1136/annrheumdis-2011-200976. Epub 2012 Mar 2. PMID 22387729
- [Background] Glazebrook KN, Kakar S, Ida CM, Laurini JA, Moder KG, Leng S. False-negative dual-energy computed tomography in a patient with acute gout. J Clin Rheumatol. 2012 Apr;18(3):138-41. doi: 10.1097/RHU.0b013e318253aa5e. PMID 22426590
- [Background] Huppertz A, Hermann KG, Diekhoff T, Wagner M, Hamm B, Schmidt WA. Systemic staging for urate crystal deposits with dual-energy CT and ultrasound in patients with suspected gout. Rheumatol Int. 2014 Jun;34(6):763-71. doi: 10.1007/s00296-014-2979-1. Epub 2014 Mar 12. PMID 24619560
- [Background] Bongartz T, Glazebrook KN, Kavros SJ, Murthy NS, Merry SP, Franz WB 3rd, Michet CJ, Veetil BM, Davis JM 3rd, Mason TG 2nd, Warrington KJ, Ytterberg SR, Matteson EL, Crowson CS, Leng S, McCollough CH. Dual-energy CT for the diagnosis of gout: an accuracy and diagnostic yield study. Ann Rheum Dis. 2015 Jun;74(6):1072-7. doi: 10.1136/annrheumdis-2013-205095. Epub 2014 Mar 25. PMID 24671771
- [Background] Jia E, Zhu J, Huang W, Chen X, Li J. Dual-energy computed tomography has limited diagnostic sensitivity for short-term gout. Clin Rheumatol. 2018 Mar;37(3):773-777. doi: 10.1007/s10067-017-3753-z. Epub 2017 Aug 12. PMID 28803339
- See also: Information about the study for patients and treating physicians in German — https://www.copago-studie.de/